CLINICAL TRIAL: NCT06441240
Title: Evaluation of Recurrence Risk Factors in Locally Advanced Breast Cancer Patients Underwent Neoadjuvant Chemotherapy. The NEORISK Study.
Brief Title: Evaluation of Recurrence Risk Factors in Locally Advanced Breast Cancer Patients Underwent Neoadjuvant Chemotherapy.
Acronym: NEORISK
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 6081
Record Dates: First submitted 2024-04-29; First posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-04

CONDITIONS: Breast Cancer; Chemotherapy Effect; Triple Negative Breast Cancer; Recurrence, Local Neoplasm; Risk Factors
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms; Neoplasm Recurrence, Local

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Breast cancer patients underwent neoadjuvant chemotherapy: Patients undergoing neoadjuvant chemotherapy and subsequent surgical treatment. Patients must have undergone radiological evaluation by MRI at the beginning and end of chemotherapy treatment
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — Breast MRI

SUMMARY:
INTRODUCTION Breast cancer (BC) is the leading cause of cancer-related death in women. Since the early 1980s, the implementation of screening programs has reduced the number of patients diagnosed with locally advanced breast cancer. Currently, the treatment for these patients involves initial neoadjuvant chemotherapy (NACT) followed by surgical treatment. In recent years, NACT has also been used for highly chemoresponsive tumors such as triple-negative (TN) and HER2-positive (HER2+) breast cancer.

The widespread use of NACT has led to additional benefits, including downstaging of breast and axillary neoplasms, resulting in reduced morbidity; improved cosmetic outcomes due to increased use of conservative interventions; and personalized adjuvant chemotherapy treatment. Several studies have shown that response to chemotherapy predicts better systemic outcomes. Complete pathological response (pCR), defined as the absence of invasive neoplastic residue in the surgical specimen, has been predictive of better distant outcomes. Limited evidence exists regarding other predictive factors for distant outcomes.

Given the significant impact of disease recurrence on patient prognosis, efforts have been made to understand the factors contributing to recurrence and to predict which patients are more prone to relapse. In this context, the term "Early Disease Recurrence" (EDR) has been coined to define the occurrence of disease recurrence, both locally and distantly, within 3 years after completing treatment.

In recent years, the potential of radiomic analysis in aiding diagnostic and therapeutic decision-making processes in BC has been demonstrated. Specifically, radiomic features obtained from Magnetic Resonance Imaging (MRI) images appear capable of predicting tumor receptor status, differentiating tumor subtypes, and predicting response to NACT.

Although the role of radiomics in predicting recurrence has been investigated, research is still in its early stages, and there are variations in technology and methodology for extracting radiomic features. Additionally, to date, no studies have evaluated the feasibility and reliability of using radiomic models combined with clinical and radiological variables to predict disease recurrence in BC patients undergoing NACT.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of locally advanced Luminal or HER2+ or Triple-negative breast cancer (cT2, T3, T4 N0 or any T N1, N2, N3, M0), clinical stage of disease from I to III.
* Patient undergoing neoadjuvant chemotherapy treatment from January 1, 2014, to June 30, 2021.
* Age > 18 years
* Availability of clinical data, staging MRI diagnostic images (for the radiomic sub-study), and biomolecular data.

Exclusion Criteria:

* Previous or synchronous history of systemic malignancies.
* History of ipsilateral or contralateral breast neoplasia.
* Evidence of metastatic disease (Stage IV).
* Neoadjuvant treatment with hormone therapy.
* Patients with unavailable or low-quality MRI images that did not allow lesion identification (for the radiomic study only).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with breast cancer (Stage I, II, and III) undergoing NACT at our center between January 2014 and June 2021 will be included, for an estimated total of 933 patients.
Sampling Method: Probability Sample
Enrollment: 933 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Description of molecular subtypes | 7 years
  Frequency of molecular subtypes (Her2 positive, hormone receptor-positive/Her2 negative, Triple Negative) in the considered cases
Association between radiomic features and risk of recurrence | 7 years
  Association between radiomic features extracted from pre-operative MRI and the onset of disease recurrence within 3 years from the end of neoadjuvant treatment

SECONDARY OUTCOMES:
Association between chemotherapy and neoplastic characteristics | 7 years
  Evaluate whether clinical features (divided into: age assessed in years, menopausal status divided into menopausal or fertile age), radiological features such as initial extent of disease and lymph node involvement at diagnosis) and biomolecular features (such as histotype: divided into ductal, lobular or nonspecial type, grading, hormone receptor status) influence response to neoadjuvant chemotherapy
  Translated with DeepL.com (free version)
Evaluation of radiological response | 7 years
  Frequency of radiological response according to molecular subtype, treatment, type of imaging examination used, and initial staging.
Frequency of complete pathological response | 7 years
  Frequency of complete pathological response according to molecular subtype, treatment, and initial staging.
Description of surgical treatment according to the cancer characteristics | 7 years
  Frequency of surgical procedures based on radiological response, molecular subtypes, and initial staging.
Description of adjuvant treatments | 7 years
  Frequency of adjuvant therapies based on neoadjuvant treatment, molecular subtypes, and initial staging.
Evaluation of oncological outcomes | 7 years
  Disease-free survival (DFS) measured from the start of neoadjuvant therapy to the first evidence of disease recurrence or death, whichever occurs first.
Assessment of risk of recurrence using models | 7 years
  Accuracy of pure models (radiomic/clinical/radiological) and combined models in predicting disease recurrence within 3 years from the end of neoadjuvant treatment

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Fabi, Principal Investigator — Policlinico Gemelli
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli - IRCCS, Roma, Italy

REFERENCES:
- [Derived] Antonio F, Carbognin L, Paris I, Di Leone A, Orlandi A, Marazzi F, Mule A, Belli P, Rossi A, Magno S, Palazzo A, Masiello V, Santoro A, Fuso P, Bria E, D'Archi S, Scardina L, Sanchez AM, Giannarelli D, Paternello S, Garganese G, Scambia G, Tortora G, Masetti R, Franceschini G, Fabi A. Predictive risk factors of recurrence in breast cancer after neoadjuvant treatment: the NEORISK study. Future Oncol. 2025 Jul;21(17):2215-2223. doi: 10.1080/14796694.2025.2516410. Epub 2025 Jun 14. PMID 40515524